CLINICAL TRIAL: NCT06058741
Title: Venetoclax Real-World Observational Study on Effectiveness and Treatment Management in Patients With Newly Diagnosed AML Who Are Ineligible for Intensive Chemotherapy in Italy
Brief Title: A Study to Asses Effectiveness and Treatment Management of Oral Venetoclax Tablets + Subcutaneously Injected Azacitidine in Adult Participants Ineligible for Intensive Chemotherapy With de Novo Acute Myeloid Leukemia (AML) in Italy
Acronym: VERO
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-498
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Venetoclax; Venclexta; Venclyxto; Azacitidine; ABT-199; Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax + Azacitidine Participants: Participants treated with venetoclax in combination with azacitidine in accordance with approved local label.

SUMMARY:
Acute myeloid leukemia (AML) is a cancer of the blood and bone marrow and is the most common acute leukemia in adults. This study will evaluate how well venetoclax in combination with azacitidine works to treat AML in newly diagnosed adult participants who are ineligible for intensive chemotherapy in Italy.

Venetoclax in combination with azacitidine is approved in Italy to treat Acute myeloid leukemia (AML) in newly diagnosed adults who are ineligible for intensive chemotherapy. All study participants will receive venetoclax in combination with azacitidine as prescribed by their study doctor in accordance with approved local label. Adult participants with a new diagnosis of AML will be enrolled. Around 150 participants will be enrolled in the study at approximately 20-25 sites in Italy.

Participants will receive venetoclax tablets to be taken by mouth in combination with azacitidine given by subcutaneous (SC) injection according to the approved local label. The duration of the study is approximately 18 months.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice and participants will be followed for 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary or secondary acute myeloid leukemia (AML), deemed ineligible for intensive induction chemotherapy because of age, performance status, comorbidities or any other clinical reason as defined by the treating physician.
* Investigator decision on patient treatment with venetoclax + azacitidine must have been reached prior to and independently of recruitment in the study.
* Treatment prescribed in accordance with the applicable approved label and local regulatory and reimbursement policies.

Exclusion Criteria:

* Participants affected by Acute Promyelocytic Leukemia.
* Prior treatment for AML, excluding hydroxyurea.
* Participation in a clinical trial of an investigational drug, concurrently or within the last 30 days. Participation in another post-marketing observational study or Registry is acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed AML participants who are ineligible to intensive chemotherapy, that starting treatment with Venetoclax in combination with azacitadine treated according to the Italian label.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 18 Months
  OS is defined as time from treatment initiation to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (28):
- Italy (28):
  - Presidio Ospedaliero Vito Fazzi /ID# 261222, Lecce, Apulia
  - Azienda Ospedaliero Universitaria Careggi /ID# 259766, Florence, Firenze
  - Ospedale San Martino /ID# 258981, Genoa, Genova
  - IRCCS Istituto Clinico Humanitas /ID# 259300, Rozzano, Lombardy
  - ASST Valle Olona/Ospedale di Busto Arsizio /ID# 259833, Busto Arsizio, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 259455, Milan, Milano
  - Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli /ID# 261794, Naples, Napoli
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 258720, Turin, Piedmont
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 260963, Meldola, Reggio Emilia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 260683, Rome, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 260821, Rome, Roma
  - AST Pesaro Urbino /ID# 261400, Pesaro, The Marches
  - Azienda Ospedaliero Universitaria delle Marche /ID# 261822, Ancona
  - ASST Papa Giovanni XXIII /ID# 258727, Bergamo
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 259535, Bologna
  - AOU Policlinico G. Rodolico - San Marco /ID# 261223, Catania
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 260738, Milan
  - Azienda Ospedaliero-Universitaria di Modena /ID# 259189, Modena
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 259778, Novara
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 261146, Palermo
  - Fondazione IRCCS Policlinico San Matteo /ID# 259624, Pavia
  - Azienda Ospedaliera di Perugia - Ospedale S. Maria della Misericordia /ID# 258983, Perugia
  - Azienda Sanitaria Locale Pescara-Presidio Ospedaliero S.Spirito /ID# 261304, Pescara
  - Grande Ospedale Metropolitano Bianchi - Melacrino - Morelli P.O. Riuniti /ID# 260737, Reggio Calabria
  - AOU San Giovanni di Dio Ruggi d'Aragona - Scuola Medica Salernitana /ID# 259456, Salerno
  - Azienda Sanitaria Universitaria Giuliano Isontina /ID# 261298, Trieste
  - Azienda Ospedaliera Universitaria Integrata di Verona /ID# 260809, Verona
  - Ospedale Belcolle /ID# 259563, Viterbo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P23-498